CLINICAL TRIAL: NCT03867123
Title: A Phase 1B Study of the Safety of LAM561 Administered Orally in Combination With Temozolomide (TMZ) and Radiation Therapy or With TMZ Alone in the First Line Treatment of Subjects With Glioblastoma
Brief Title: A Study to Evaluate the Safety of LAM561 Added to Standard of Care in Newly-diagnosed Glioblastoma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laminar Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIN-002-1801; 2018-000317-21 (EudraCT Number)
Record Dates: First submitted 2019-01-03; First posted 2019-03-07 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Glioblastoma (GBM)
MeSH Terms: conditions — Glioblastoma | interventions — Radiotherapy; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (chemoradiation phase) (Experimental): Radiotherapy (RT) + temozolomide (TMZ) + LAM561 (during Concurrent phase - duration 6 weeks)*:
  LAM561 will be initiated at the start of the concurrent phase and will be administered on a continuous daily basis together with TMZ and RT for 6 weeks at the selected dose, either 12 g/day (4 g tid), 8 g/day (4 g bid) or 4 g/day (4 g od).
  RT will be administered only during the concurrent phase, consisting of fractionated focal irradiation administered using 1.8- 2 Gy/fraction, daily for 5 days/week for 6 weeks, for a total dose of up to 60 Gy.
  TMZ will be administered during the concurrent phase at a starting dose of 75 mg/m2/day given daily for 6 weeks.
  * One extra week may be allowed.
  Interventions: Drug: LAM561; Radiation: RT; Drug: TMZ
- Arm 2 (maintenance phase) (Experimental): TMZ + LAM561 (during Maintenance phase with TMZ 200 mg/m2/day at Cycle 2 - duration 8 weeks):
  LAM561 will be initiated on day 2 of Cycle 2 of the maintenance phase, when TMZ 200 mg/m2/day is given and administered on a continuous basis for two 28-day cycles. LAM561 will be administered at the selected dose, either 12 g/day (4 g tid), 8 g/day (4 g bid) or 4 g/day (4 g od).
  TMZ will be administered at 200 mg/m2/day given daily the first 5 days for two 28-day cycles (if no toxicity is seen). In case of toxicity, TMZ dose may be reduced to 150 mg/m2/day at Cycle 3 to allow for recovery.
  Both arms will be followed by a 4-week safety follow-up
  Interventions: Drug: LAM561; Drug: TMZ

INTERVENTIONS:
Drug: LAM561 — Arm 1: Daily for 6 weeks. Arm 2: daily, two 28-day cycles
Radiation: RT — In Arm 1: Fractionated focal irradiation of 1.8-2 Gy/fraction/day, 5 days/week, 6 weeks. Total dose up to 60 Gy
  Other Names: radiotherapy
  Arms: Arm 1 (chemoradiation phase)
Drug: TMZ — Arm 1: 75 mg/m2/day, daily, 6 weeks Arm 2: 200 mg/m2/day, daily the first 5 days of two 28-day cycles (in case of toxicity, TMZ dose may be reduced to 150 mg/m2/day at Cycle 3 to allow for recovery)
  Other Names: temozolomide

SUMMARY:
The purpose of this study is to determine the safety and tolerability of LAM561 added to first-line treatment for subjects with newly diagnosed glioblastoma (GBM), and to determine the highest safe dose of LAM561 administered orally when added to the concurrent phase of treatment with temozolomide (TMZ) and radiation therapy (RT) or when added to the maintenance phase of treatment with TMZ (once TMZ 200 g/m2/day is started).

DETAILED DESCRIPTION:
This is a Phase IB, open-label, dose-finding study. A de-escalation process has been selected for the study with a 3+3 design to establish the Maximum Tolerated Dose (MTD).

The first group of 3 subjects (within each arm), where all 3 subjects may be started at the same time, will receive LAM561 at the starting dose of 12 g/day (4 g tid). If 0-1 Dose-Limiting Toxicities (DLTs) in the first 3 patients, then a new cohort with 3 more patients is started at 12 g/day (4 g tid). If 2 or more patients out of 3 or 6 patients experience DLT(s) the dose is deescalated.

De-escalation doses are from 12 g/day (4 g tid) to 8 g/day (4 g bid) and from 8 g/day (4 g bid) to 4 g/day (4 g od). This procedure must be applied to the two arms of the study described below. Both arms will be independent, and will run in parallel, therefore none of the patients from Arm 1 may enter Arm 2.

ELIGIBILITY:
Inclusion Criteria:

1. Glioblastoma (GBM) according to 2016 World Health Organization (WHO) Classification.
2. Must have had a partial or complete surgical resection of the Grade 4 astrocytic tumor.
3. Subjects in Arm 1 must have had no previous treatment except surgery (ie, no previous RT, local CT, or systemic therapy). Subjects must meet certain other eligibility requirements.
4. Subjects in Arm 2 must have completed a standard first line regimen of concurrent TMZ and RT for newly diagnosed GBM patients, followed by a rest phase, and have not had any other previous CT except surgery (including any other regimens of RT and local or systemic CT). Progression and/or pseudoprogression should have been ruled out before starting Arm 2 as per usual clinical practice, with correct laboratory results (absolute neutrophile count ≥1.5 x 109/L, platelet count ≥ 100 x 109/L, non-haematological toxicity grade ≤ 2) at screening. Subjects must meet certain other eligibility requirements.
5. Subjects must be able to undergo serial MRIs (computerized tomography may not be a substitute for magnetic resonance imaging [MRI]).
6. Male or female ≥ 18 years old.
7. Must have a Karnofsky performance status of ≥ 70% and the ability to swallow oral medication.
8. Must have no other diagnosis of cancer malignancy (except surgically excised nonmelanoma skin cancer or carcinoma in situ of the cervix, or treated early stage prostate cancer, or a malignancy diagnosed ≥ 5 years previously with no current evidence of disease and no therapy within two years prior to enrolment on this study).
9. Must be capable of understanding and complying with the protocol requirements.
10. Contraception: All female patients will be considered to be of childbearing potential unless they are postmenopausal (at least 12 months consecutive amenorrhea, in the appropriate age group and without other known or suspected cause), or have been sterilized surgically. Female patients of childbearing potential must agree to use two forms of highly effective contraception methods (a primary and a secondary method) during the study and for a period of 6 months following the last administration of the study drug. Male patients and their female partners, who are of childbearing potential and are not practicing total abstinence, must agree to use two forms of highly effective contraception methods (a primary and a secondary method) during the study and for a period of 6 months following the last administration of the study drug These contraception methods include oral, transdermal, systemic or implant contraception birth control, intra-uterine devices (IUD), abstinence and double barrier method such as diaphragm with spermicidal gel or other recommended double barrier methods screening.
11. Written informed consent form signed before any study test or procedure.

Exclusion Criteria:

1. Subject has received prior systemic CT or RT (Arm 1) or prior systemic CT other than TMZ (Arm 2), biologic agents, or any other type of investigational agent for the treatment of brain tumors.
2. Subjects who have progressed on TMZ are not eligible (pseudoprogression ruled out as per usual clinical practice).
3. Subject has evidence of acute intracranial or intratumoral hemorrhage > Grade 1 by MRI. Subjects with resolving hemorrhage changes, punctate hemorrhage, or hemosiderin may enter the study.
4. Subject has serious intercurrent illness such as: hypertension despite optimal treatment, or significant cardiac arrhythmias; or a recent history of serious disease such as symptomatic congestive heart failure, or abdominal fistula or gastrointestinal (GI) perforation within 6 months, prior to starting study treatment.
5. Subject has had major surgery within 28 days prior to starting study treatment (except cancer resection surgery in arm 1), or had non water-tight dural closure during previous surgery, or has unhealed wounds from previous surgery.
6. Subject has inherited bleeding diathesis or coagulopathy with the risk of bleeding.
7. Subject is pregnant or breastfeeding.
8. Subject is known to be positive for the human immunodeficiency virus (HIV) (a test for HIV at screening is not required).
9. Subject has a previously-identified allergy or hypersensitivity to components of either the LAM561 or TMZ formulations.
10. Subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of LAM561 in association with Standard of Care (Stupp Protocol) | 10 to 12 weeks
  Incidence of Treatment-Emergent Adverse Events.
Maximum Tolerated dose (MTD) | 10 to 12 months
  MTD of LAM561 administered with Standard of Care

SECONDARY OUTCOMES:
Plasma concentration of temozolomide (TMZ). | First five days of cycle 2 of maintenance phase (each cycle is 4 weeks)
  To verify that the administration of LAM561 is not modifying the exposition of patients to TMZ.

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Roma, MD, Study Director — cro
Locations (3):
- Spain (3):
  - Institut Catala d'Oncologia, Hospital Germans Trias I Pujol, Badalona, Catalonia
  - Hospital Universitari de Girona Dr. Josep Trueta, Institut Català d'Oncologia, Girona, Catalonia
  - Hospital Duran i Reynals, Institut Català d'Oncologia, L'Hospitalet de Llobregat, Catalonia

IPD SHARING:
Plan to Share IPD: Undecided